CLINICAL TRIAL: NCT02499380
Title: Changes in Lung Physiology and Cardiac Performance in Patients With Emphysema Post Bilateral RePneu Coil Treatment
Status: Terminated | Type: Observational
Why Stopped: Study enrollment was prematurely stopped.
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0017
Record Dates: First submitted 2015-05-27; First posted 2015-07-16 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: RePneu; Coil; LVRC; PneumRx
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Patients treated with PneumRx Coil System
  Interventions: Device: PneumRx Coil System

INTERVENTIONS:
Device: PneumRx Coil System
  Other Names: LVRC; RePneu

SUMMARY:
The objective of this post-marketing study is to advance the understanding of the mechanism of action of the CE marked RePneu Coil by observing changes in lung physiology and cardiac performance in patients with emphysema treated with the RePneu Coils, when used as intended.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects diagnosed with emphysematous type of COPD.
2. CT scan indicates bilateral emphysema, with sufficient lung parenchyma for coil deployment (based on PneumRx CT scoring) criteria.
3. Subject has post-bronchodilator FEV1 ≤45% predicted.
4. Subject has Total Lung Capacity >100% predicted.
5. Subject has residual volume (RV) ≥175% predicted.
6. Subject has marked dyspnea scoring ≥2 on mMRC scale of 0-4.
7. Subject read, understood and signed the Informed Consent form.
8. Subject has received Pneumococcal and Influenza vaccinations consistent with local recommendations and/or policy.

Exclusion Criteria:

1. Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g. severe arthritis, planned knee surgery) or baseline limitation not due to dyspnea.
2. Subject has a change in FEV1 >20% (or, for subjects with pre-bronchodilator FEV1 below 1 L, a change of > 200 mL) post-bronchodilator unless investigator can confirm by other means that subject does not have asthma.
3. Subject has severe gas exchange abnormalities as defined by:

   * PaCO2 >55 mm Hg
   * PaO2 <45 mm Hg on room air (High altitude criterion: PaO2 <30 mm Hg)
4. Subject has severe pulmonary hypertension defined by right ventricular systolic pressure >50 mm Hg via right heart catheterization and/or echocardiogram.
5. Subject has evidence of other severe disease (such as, but not limited to, lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
6. Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
7. Subject has an inability to tolerate bronchoscopy under moderate sedation or general anesthesia.
8. Subject has clinically significant bronchiectasis.
9. Subject has had previous LVR surgery, lung transplantation, lobectomy or other BLVR treatment in either lung.
10. Subject has participated in studies to treat COPD using high dose radiation.
11. Subject has been involved in pulmonary drug or device studies within 30 days prior to this study.
12. Subject is chronically taking >20 mg prednisone (or equivalent dose of a similar steroid) daily.
13. Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
14. Subject is on any type of antiplatelet or anticoagulant therapy which cannot be stopped for seven (7) days prior to procedure.
15. Subject has a sensitivity or allergy to Nickel.
16. Subject has a known sensitivity to drugs required to perform bronchoscopy.
17. Subject has been diagnosed with alpha-1 antitrypsin deficiency (AATD).
18. Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow-up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects diagnosed with emphysematous type of COPD
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Lungenclinic, Großhansdorf
  - Thoraxklinik, Heidelberg

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients treated with PneumRx Coil System
  PneumRx Coil System
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.50 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in 6 Minute Walk Distance (6MWD)
Description: Changes in distance traveled during a 6 minute walk test (6MWT). Initial baseline measurement was taken prior to the treatment with the RePneu coil and the second measurement was taken 12 months after the initial treatment of the RePneu coil. 6MWD was measured in meters.
Time Frame: Baseline, 12 months post initial treatment
Population: Intention to treat population with 6MWT data available at baseline and 12 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment
Number analyzed (Participants) | 15
meters | 19.1 (63.06)

2. Primary Outcome: Changes in 6 Minute Walk Distance (6MWD)
Description: Changes in distance traveled during a 6 minute walk test (6MWT). Initial baseline measurement was taken prior to the treatment with the RePneu coil and the second measurement was taken 3 months after final treatment of the RePneu coil. 6MWD was measured in meters.
Time Frame: Baseline, 3 months post final treatment
Population: Intention to treat population with 6MWT data available at baseline and 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment
Number analyzed (Participants) | 14
meters | 21.4 (46.94)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Condition aggravated (General disorders) | 1 (1)
Implant site reaction (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Infective exacerbation of chronic obstructive pulmonary disorders (Infections and infestations) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
General Physical Health Deterioration (General disorders) | 1 (1)
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Mastectomy (Surgical and medical procedures) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-08-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02499380/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02499380/SAP_001.pdf